CLINICAL TRIAL: NCT06496178
Title: A Phase 3 Open-label, Randomized Controlled Study to Evaluate the Efficacy and Safety of Petosemtamab Compared With Investigator's Choice Monotherapy Treatment in Previously Treated Patients With Incurable, Metastatic/Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: A Phase 3 Study to Evaluate Petosemtamab Compared With Investigator's Choice Monotherapy in Previously Treated Head and Neck Squamous Cell Carcinoma Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-158-CL02; 2023-510322-32 (EudraCT Number)
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MCLA-158 (Experimental)
  Interventions: Drug: Petosemtamab
- Investigator's Choice (Active Comparator)
  Interventions: Drug: Investigator's Choice

INTERVENTIONS:
Drug: Petosemtamab — MCLA-158
  Arms: MCLA-158
Drug: Investigator's Choice — Cetuximab
  Arms: Investigator's Choice
Drug: Investigator's Choice — Methotrexate
  Arms: Investigator's Choice
Drug: Investigator's Choice — Docetaxel
  Arms: Investigator's Choice

SUMMARY:
This is a phase 3 open-label, randomized, controlled, multicenter study to compare petosemtamab vs investigator's choice monotherapy in HNSCC patients for the second- and third-line treatment of incurable metastatic/recurrent disease.

DETAILED DESCRIPTION:
This is a phase 3 open-label, randomized, controlled, multicenter study to compare petosemtamab vs investigator's choice monotherapy in HNSCC patients for the second- and third-line treatment of incurable metastatic/recurrent disease. HNSCC patients must have progressive disease (PD) on or after anti-PD-1 therapy and platinum-containing therapy. Patients treated with platinum-containing therapy only in the adjuvant setting, or in the context of multimodal therapy for locally advanced disease, should have PD within 6 months of the last dose of platinum-containing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF before initiation of any study procedures.
* Age ≥ 18 years at signing of ICF.
* Histologically previously confirmed HNSCC with evidence of metastatic or locally advanced disease not amenable to standard therapy with curative intent.
* HNSCC patients progressed on or after anti-PD-1 therapy and platinum-containing therapy.
* The eligible HNSCC primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
* Documentation of p16 status (positive or negative) by local laboratory IHC for patients with primary oropharyngeal cancer.
* A baseline new tumor sample unless the patient has an available tumor sample as an FFPE block with sufficient material.
* Measurable disease as defined by RECIST v1.1 by radiologic methods.
* ECOG PS of 0 or 1
* Life expectancy ≥ 12 weeks, as per investigator
* Adequate organ function (as per protocol)

Exclusion Criteria:

* Central nervous system metastases that are untreated or symptomatic, or require radiation, surgery, or continued steroid therapy to control symptoms within 14 days of study entry.
* Known leptomeningeal involvement
* Any systemic anticancer therapy within 4 weeks of the first dose of study treatment.
* Major surgery or radiotherapy within 3 weeks of the first dose of study treatment.
* Persistent Grade >1 clinically significant toxicities related to prior antineoplastic therapies
* History of hypersensitivity reaction to any of the excipients of treatment required for this study.
* Unstable angina; history of congestive heart failure of Class II-IV New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment or history of myocardial infarction within 6 months of study entry
* History of prior malignancies with the exception of excised cervical intraepithelial neoplasia or nonmelanoma skin cancer, or curatively treated cancer deemed at low risk for recurrence with no evidence of disease
* Current dyspnea at rest of any origin, or other diseases requiring continuous oxygen therapy
* Current serious illness or medical conditions including, but not limited to, uncontrolled active infection, clinically significant pulmonary, metabolic or psychiatric disorders
* Patients with known infectious diseases (as per protocol)
* Pregnant or breastfeeding patients
* Patient has a primary tumor site of nasopharynx (any histology).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review | Up to approximately 2 years
  ORR was defined as the proportion of participants in the analysis population who had a Complete Response or Partial Response based per RECIST v1.1 with confirmation.
Overall Survival (OS) | Up to approximately 3 years
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) as Assessed by Blinded Independent Central Review | Up to approximately 2 years
  PFS was defined as the time from randomization to the first documented disease progression per RECIST v1.1 or death due to any cause.
Duration of Response (DOR) as Assessed by Blinded Independent Central Review | Up to approximately 2 years
  For participants with a confirmed CR or PR per RECIST v1.1, DOR was defined as the time from the date of first documented response of CR or PR per RECIST v1.1 to the date of first documented progression or death due to underlying cancer.
Objective Response Rate (ORR) as Assessed by Investigator Review | Up to approximately 2 years
  ORR was defined as the proportion of participants in the analysis population who had a Complete Response or Partial Response based per RECIST v1.1 with confirmation.
Progression Free Survival (PFS) as Assessed by Investigator Review | Up to approximately 2 years
  PFS was defined as the time from randomization to the first documented disease progression per RECIST v1.1 or death due to any cause.
Duration of Response (DOR) as Assessed by Investigator Review | Up to approximately 2 years
  For participants with a confirmed CR or PR per RECIST v1.1, DOR was defined as the time from the date of the first documented response of CR or PR per RECIST v1.1 to the date of first documented progression or death due to underlying cancer.
Time to Response (TTR) as Assessed by Blinded Independent Central Review | Up to approximately 2 years
  For participants with a confirmed CR or PR per RECIST v1.1, TTR was defined as the time from randomization to the first documented response per RECIST v1.1.
Time to Response (TTR) as Assessed by Investigator Review | Up to approximately 2 years
  For participants with a confirmed CR or PR per RECIST v1.1, TTR was defined as the time from randomization to the first documented response per RECIST v1.1.
Clinical Benefit Rate (CBR) as Assessed by Blinded Independent Central Review | Up to approximately 2 years
  CBR was defined as the proportion of participants with a confirmed CR or PR, or SD lasting 16 weeks for longer per RECIST v1.1
Clinical Benefit Rate (CBR) as Assessed by Investigator Review | Up to approximately 2 years
  CBR was defined as the proportion of participants with a confirmed CR or PR, or SD lasting 16 weeks for longer per RECIST v1.1
Number of participants Who experienced At Least One Treatment Emergent Adverse Event (TEAE) | Up to 30 days post-last dose
  An AE means any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related. The term TEAE covers any unfavorable and unintended sign, symptom, syndrome, or illness that develops or worsens during the period of observation after the first treatment administration in the clinical study. The number of all participants who experienced at least one TEAE is presented.
Number of participants Who experienced At Least One Serious TEAE | Up to 30 days post-last dose
  An AE means any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related. The term TEAE covers any unfavorable and unintended sign, symptom, syndrome, or illness that develops or worsens during the period of observation after the first treatment administration in the clinical study. The number of all participants who experienced at least one serious TEAE is presented.
Number of participants Who Discontinued Study Treatment Due to TEAEs | Up to 30 days post-last dose
  An AE means any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related. The term TEAE covers any unfavorable and unintended sign, symptom, syndrome, or illness that develops or worsens during the period of observation after the first treatment administration in the clinical study. The number of all participants who discontinued study treatment due to TEAEs is presented.
Number of participants Who Had Dose Modification Due to TEAEs | Up to 30 days post-last dose
  An AE means any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related. The term TEAE covers any unfavorable and unintended sign, symptom, syndrome, or illness that develops or worsens during the period of observation after the first treatment administration in the clinical study. The number of all participants who had dose modification due to TEAEs is presented.
Mean Change From Baseline in EORTC QLQ-C30 | Up to approximately 2 years
  For the EORTC QLQ-C30, the functional scales, the symptom scales, the specific single items, and the global health and quality of life scale, will be computed according to EORTC QLQ-C30 Scoring Manual. Mean change from baseline is presented.
Mean Change From Baseline in EORTC QLQ-H&N43 | Up to approximately 2 years
  For the updated EORTC QLQ-H&N43, the multi-item scales and the single-items will be computed according to EORTC QLW-HN43 Scoring Manual. Mean change from baseline is presented.
Concentrations Predose And at End of Infusion | Up to first 6 cycles
  Predose and end of infusion plasma concentrations as measured from all individual plasma concentrations.
Pharmacokinetic parameters | Up to first 6 cycles
  Clearance of plasma and central volume of distribution based on population PK model
Incidence of anti-drug antibody (ADA) | Up to 30 days post-last dose
  The frequency and proportion of participants developing anti-drug antibodies.

CONTACTS AND LOCATIONS:
Locations (197):
- United States (57):
  - Site 160, Mobile, Alabama
  - Site 102, Prescott, Arizona
  - Site 125, Scottsdale, Arizona
  - Site 82, Duarte, California
  - Site 25, La Jolla, California
  - Site 173, Orange, California
  - Site 28, Palo Alto, California
  - Site 127, Sacramento, California
  - Site 46, San Francisco, California
  - Site 130, Lone Tree, Colorado
  - Site 104, Washington D.C., District of Columbia
  - Site 12, Fort Myers, Florida
  - Site 123, Jacksonville, Florida
  - Site 9, Orlando, Florida
  - Site 138, Temple Terrace, Florida
  - Site 187, Atlanta, Georgia
  - Site 152, Chicago, Illinois
  - Site 68, Chicago, Illinois
  - Site 31, Indianapolis, Indiana
  - Site 8, Louisville, Kentucky
  - Site 40, Baton Rouge, Louisiana
  - Site 100, New Orleans, Louisiana
  - Site 153, Columbia, Maryland
  - Site 77, Boston, Massachusetts
  - Site 103, Ann Arbor, Michigan
  - Site 5, Detroit, Michigan
  - Site 49, Maple Grove, Minnesota
  - Site 124, Rochester, Minnesota
  - Site 18, St Louis, Missouri
  - Site 86, Hackensack, New Jersey
  - Site 15, Albuquerque, New Mexico
  - Site 24, New York, New York
  - Site 98, Chapel Hill, North Carolina
  - Site 122, Durham, North Carolina
  - Site 23, Cincinnati, Ohio
  - Site 87, Cleveland, Ohio
  - Site 32, Columbus, Ohio
  - Site 26, Portland, Oregon
  - Site 151, Bensalem, Pennsylvania
  - Site 158, Philadelphia, Pennsylvania
  - Site 159, Philadelphia, Pennsylvania
  - Site 50, Charleston, South Carolina
  - Site 60, Chattanooga, Tennessee
  - Site 54, Memphis, Tennessee
  - Site 59, Nashville, Tennessee
  - Site 67, Nashville, Tennessee
  - Site 55, Denison, Texas
  - Site 34, El Paso, Texas
  - Site 51, Houston, Texas
  - Site 7, Houston, Texas
  - Site 94, Pearland, Texas
  - Site 4, Salt Lake City, Utah
  - Site 10, Blacksburg, Virginia
  - Site 22, Charlottesville, Virginia
  - Site 156, Winchester, Virginia
  - Site 163, Seattle, Washington
  - Site 6, Spokane, Washington
- Argentina (7):
  - Site 37, Buenos Aires
  - Site 80, Buenos Aires
  - Site 58, Caba
  - Site 193, CABA
  - Site 45, Córdoba
  - Site 110, Rosario
  - Site 57, Viedma
- Australia (6):
  - Site 3, Darlinghurst
  - Site 170, Herston
  - Site 38, Melbourne
  - Site 30, Nedlands
  - Site 11, Saint Leonards
  - Site 73, Sydney
- Belgium (6):
  - Site 129, Brussels
  - Site 56, Brussels
  - Site 92, Ghent
  - Site 72, Leuven
  - Site 108, Liège
  - Site 69, Namur
- Brazil (8):
  - Site 154, Brasília
  - Site 145, Porto Alegre
  - Site 150, Porto Alegre
  - Site 146, Recife
  - Site 155, Rio de Janeiro
  - Site 148, Rio de Janeiro
  - Site 147, São Paulo
  - Site 144, São Paulo
- Canada (2):
  - Site 172, Montreal
  - Site 196, Toronto
- Chile (4):
  - Site 16, Providencia
  - Site 20, Recoleta
  - Site 27, Santiago
  - Site 21, Santiago
- Site 188, Nový Jičín, Czechia
- France (15):
  - Site 105, Bordeaux
  - Site 162, Le Mans
  - Site 149, Lille
  - Site 118, Lyon
  - Site 115, Marseille
  - Site 106, Montpellier
  - Site 169, Nice
  - Site 114, Paris
  - Site 167, Paris
  - Site 136, Poitiers
  - Site 141, Rennes
  - Site 107, Rouen
  - Site 119, Toulouse
  - Site 142, Vandœuvre-lès-Nancy
  - Site 113, Villejuif
- Germany (12):
  - Site 101, Aachen
  - Site 121, Berlin
  - Site 165, Essen
  - Site 84, Giessen
  - Site 62, Greifswald
  - Site 79, Hamburg
  - Site 88, Hamburg
  - Site 112, Hanover
  - Site 116, Leipzig
  - Site 175, Mannheim
  - Site 168, München
  - Site 99, Würzburg
- Greece (5):
  - Site 91, Athens
  - Site 96, Athens
  - Site 120, Heraklion
  - Site 126, Rio
  - Site 83, Thessaloniki
- Site 195, Pécs, Hungary
- Israel (4):
  - Site 19, Haifa
  - Site 1, Jerusalem
  - Site 2, Tel Aviv
  - Site 14, Tel Litwinsky
- Italy (6):
  - Site 93, Brescia
  - Site 111, Cuneo
  - Site 128, Milan
  - Site 81, Milan
  - Site 89, Napoli
  - Site 85, Rozzano
- Japan (8):
  - Site 132, Chūōku
  - Site 192, Fukuoka
  - Site 131, Kashiwa
  - Site 135, Miki
  - Site 139, Nagoya
  - Site 186, Natori
  - Site 133, Ōsaka-sayama
  - Site 134, Sendai
- Lithuania (2):
  - Site 180, Kaunas
  - Site 181, Vilnius
- Netherlands (3):
  - Site 76, Amsterdam
  - Site 61, Nijmegen
  - Site 66, Utrecht
- Poland (6):
  - Site 190, Bydgoszcz
  - Site 143, Gdansk
  - Site 97, Gliwice
  - Site 177, Krakow
  - Site 117, Skorzewo
  - Site 179, Warsaw
- Portugal (4):
  - Site 182, Coimbra
  - Site 183, Lisbon
  - Site 197, Portimão
  - Site 185, Porto
- South Korea (8):
  - Site 161, Busan
  - Site 13, Goyang-si
  - Site 29, Hwasun
  - Site 137, Seoul
  - Site 36, Seoul
  - Site 47, Seoul
  - Site 33, Soeul
  - Site 164, Suwon
- Spain (8):
  - Site 78, Barcelona
  - Site 109, Madrid
  - Site 75, Madrid
  - Site 71, Madrid
  - Site 166, Madrid
  - Site 63, Pamplona
  - Site 64, Pamplona
  - Site 74, Valencia
- Switzerland (4):
  - Site 184, Bellinzona
  - Site 189, Geneva
  - Site 194, Lausanne
  - Site 178, Sankt Gallen
- Taiwan (8):
  - Site 41, Changhua
  - Site 17, Kaohsiung City
  - Site 95, Kaohsiung City
  - Site 53, Taichung
  - Site 176, Tainan
  - Site 39, Taipei
  - Site 35, Taipei
  - Site 52, Taoyuan
- United Kingdom (12):
  - Site 65, Cambridge
  - Site 174, Cardiff
  - Site 171, Glasgow
  - Site 44, Liverpool
  - Site 157, London
  - Site 140, London
  - Site 90, London
  - Site 42, London
  - Site 48, Manchester
  - Site 70, Middlesex
  - Site 191, Newcastle upon Tyne
  - Site 43, Sutton

REFERENCES:
- [Derived] Machiels JP, Fayette J, Haddad R, Adkins D, Gillison M, Harrington KJ, Kim SB, Le Tourneau C, Psyrri A, Rosenberg A, Siu LL, Tahara M, William WN Jr, Ford J, Jauhari S, Pyle R, Shen YM, Yao D, Zohren F, Vokes E. LiGeR-HN phase III trials of petosemtamab + pembrolizumab and petosemtamab monotherapy in recurrent or metastatic HNSCC. Future Oncol. 2025 Jul;21(16):2007-2016. doi: 10.1080/14796694.2025.2511470. Epub 2025 Jun 13. PMID 40511820